CLINICAL TRIAL: NCT04040959
Title: Nicotinamide Riboside Supplementation for Treating Arterial Stiffness and Elevated Systolic Blood Pressure in Patients With Moderate to Severe CKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-0149; R01DK121516-01 (NIH)
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Vascular Diseases; Kidney Disease; Blood Pressure; Oxidative Stress
Keywords: stiffness; chronic kidney disease; Hypertension
MeSH Terms: conditions — Vascular Diseases; Kidney Diseases; Renal Insufficiency, Chronic; Hypertension | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotinamide Riboside (Experimental): Each nicotinamide riboside capsule contains 250 mg of nicotinamide riboside chloride mixed with microcrystalline cellulose. Dosage: 500 mg by mouth twice a day for 3 months.
  Interventions: Drug: Nicotinamide riboside
- Placebo (Placebo Comparator): Matched placebo capsules.
  Interventions: Drug: Nicotinamide riboside

INTERVENTIONS:
Drug: Nicotinamide riboside — Nicotinamide riboside is a naturally occurring vitamin B3 derivative found in yeast, bacteria, and mammalian tissues, and also has been detected in cows' milk.

SUMMARY:
Risk of cardiovascular diseases (CVD) is significantly elevated in patients with chronic kidney disease (CKD); however, this increased risk is only partially explained by traditional CV risk factors. Arterial dysfunction is an important nontraditional CV risk factor gaining increased recognition in the field of nephrology. This process is best represented, both physiologically and pathophysiologically, by increases in the gold standard measure of arterial stiffening, carotid to femoral artery pulse wave velocity (CFPWV), which reflects, in particular, increases in aortic stiffness. Aortic stiffening with CKD is mediated by structural and functional (increased vascular smooth muscle tone) changes in the arterial wall stimulated by oxidative stress and chronic low-grade inflammation. Caloric restriction (CR) is a promising strategy for prevention of CKD-associated arterial dysfunction and CVD. However, long-term adherence to chronic CR regimens with optimal nutrition is very difficult to achieve. Research has shown that boosting NAD+ bioavailability to stimulate SIRT-1, a "CR mimetic" approach, reduces CFPW and oxidative stress in old mice, and this lab recently took the first step in translating these findings in a study of adults with normal kidney function and elevated systolic blood pressure (SBP). The data found that supplementation with nicotinamide riboside, a natural, commercially available precursor of NAD+ and novel CR mimetic, increased NAD+ bioavailability and reduced CFPWV and SBP. A randomized, placebo-controlled, double-blind, single-site phase IIa clinical trial to assess the safety and efficacy of oral nicotinamide riboside (500 mg capsules 2x/day; NIAGEN®; ChromaDex Inc.) for 3 months vs. placebo for decreasing aortic stiffness and SBP in patients (35-80 years) with stage III and IV CKD is being proposed. It is hypothesized that treatment will reduce CFPWV and SBP, as related to increases in systemic NAD+ bioavailability and reductions in oxidative stress, and inflammation.

Aim 1: To measure CFPWV (primary outcome) before/after nicotinamide riboside vs. placebo treatment; Aim 2: To measure casual and 24h-ambulatory SBP (secondary outcome) before and after treatment; Aim 3: To determine the safety and tolerability of treatment with nicotinamide riboside vs. placebo; Aim 4: To measure systemic NAD+ and NAD+-related metabolite concentrations, as well as circulating markers of oxidative stress, inflammation, and vasoconstriction factors before and after treatment.

DETAILED DESCRIPTION:
Background: Risk of cardiovascular diseases (CVD) is significantly elevated in patients with chronic kidney disease (CKD). Arterial dysfunction is an important nontraditional CV risk factor gaining increased recognition in the field of nephrology. While many changes likely contribute to the development of arterial dysfunction in patients with CKD, among those of greatest concern is the development of stiffening of the large elastic arteries. Caloric restriction (CR) is a promising strategy for prevention of CKD-associated arterial dysfunction and CVD; however, adherence to CR is poor and may be detrimental in CKD patients due to reduced skeletal muscle and bone mass. Therefore, identification of more practical interventions that mimic the beneficial effects of CR, with stronger adherence and less risk of adverse consequences, is of significant biomedical importance.

Nicotinamide riboside is a naturally occurring precursor of nicotinamide adenine dinucleotide (NAD+), a critical mediator of the beneficial effects of CR, and therefore, a novel CR mimetic compound. We recently completed a study of nicotinamide riboside supplementation in healthy middle-age and older adults and demonstrated that 6 weeks of supplementation with nicotinamide riboside lowered carotid-femoral pulse wave velocity (CFPWV), the gold-standard clinical measure of aortic stiffness and a strong independent predictor of CVD and related morbidity and mortality in patients with and without kidney disease. In addition, treatment with nicotinamide riboside decreased systolic blood pressure (SBP) by 8 mmHg compared with placebo.

As a next translational step, we propose to conduct a randomized, placebo-controlled, double-blind, single site phase IIa clinical trial to further assess the safety and efficacy of oral nicotinamide riboside (3 months vs. placebo) for decreasing aortic stiffness and SBP in patients with stage III and IV CKD. We hypothesize that nicotinamide riboside will lower aortic stiffness and SBP and that these improvements will be related to increases in systemic NAD+ bioavailability, selective influences on vascular smooth muscle tone, and reductions in markers of systemic oxidative stress and/or inflammation.

Primary Outcome Measure (Aim 1): Aortic stiffness will be evaluated as CFPWV, the gold-standard measurement technique and clinically relevant marker of vascular function. CFPWV will be measured before and after 3 months of treatment with nicotinamide riboside or placebo.

Secondary Outcome Measures (Aim 2): Casual and ambulatory SBP will be the main secondary outcomes measures: (a) Casual (resting) SBP will be measured according to American Heart Association/American College of Cardiology guidelines, with an automated oscillometric sphygmomanometer. Casual SBP will be measured before and after 3 months of treatment with nicotinamide riboside or placebo; (b) Ambulatory SBP is an independent risk factor for CVD and a predictor of target organ damage. Ambulatory SBP (24-hour, daytime, nighttime mean pressures) will be measured before and after 3 months of treatment with nicotinamide riboside or placebo.

Other Outcome Measures (Aims 3 and 4): To evaluate the safety of nicotinamide riboside, we will monitor treatment-emergent adverse events at each visit (once every 2 weeks). The most common adverse events associated with nicotinamide riboside include mild-to-moderate headache, feelings of warmth, hot flushing sensations, gastrointestinal discomfort, and fatigue. We will also evaluate safety before and after 3 months of treatment with nicotinamide riboside or placebo by measuring the following clinical markers: standard blood hematology, standard clinical chemistry profiles, and standard urinalysis.

Tolerability will be assessed as subject dropout due to treatment-emergent adverse events.

Adherence to the intervention will be assessed by pill count performed once every 2 weeks.

Concentrations of NAD+ and associated metabolites will be evaluated to determine whether oral supplementation with nicotinamide riboside increases systemic NAD+ bioavailability. Peripheral blood mononuclear cells will be isolated and quantitative targeted metabolomics will be employed to evaluate concentrations of associated metabolites.

CKD and aortic stiffness and increased blood pressure are associated with increased systemic oxidative stress, inflammation, and pro-vasoconstriction factors. Nicotinamide riboside may reduce vascular stiffness by acting on one or more of these pathways. Circulating biomarkers of potential mechanisms of action (norepinephrine, endothelin-1, C-reactive protein, oxidized low density lipoprotein, total antioxidant status, tumor necrosis factor-alpha, interleukin-6, interleukin-1 beta and interleukin-10) will be evaluated to provide mechanistic insight. All of the discussed other outcome measures will be evaluated before and after 3 months of supplementation with nicotinamide riboside or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-80 years;
* Ability to provide informed consent;
* Willing to accept random assignment to condition;
* CKD stage III or IV (eGFR with the 4-variable MDRD prediction equation: 20-60 mL/min/1.73m2; stable renal function in the past 3 months);
* Blood pressure controlled to <140/90 mmHg for the past 3 months;
* Body mass index <40 kg/m2;
* Weight stable in the prior 3 months (<2 kg weight change) and willing to remain weight stable throughout the study

Exclusion Criteria:

* Patients with advanced CKD requiring chronic dialysis;
* Significant co-morbid conditions that lead the investigator to conclude that life expectancy < 1 year;
* History of severe congestive heart failure (i.e., ejection fraction < 35%);
* Hospitalization in the past month;
* Proteinuria > 5 g/day;
* Immunosuppressant agents such as cyclosporine, tacrolimus, azathioprine, etanercept, infliximab, adalimumab, anakinra or long-term oral glucocorticoids taken in past 12 months;
* Known malignancy;
* Woman who are pregnant, nursing or planning to become pregnant;
* Special classes of subjects considered vulnerable populations will not be included in the study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
carotid-femoral pulse wave velocity | Baseline and 3 months
  change in carotid-femoral pulse wave velocity

SECONDARY OUTCOMES:
Systolic blood pressure | Baseline and 3 months
  Casual blood pressure
Systolic blood pressure | Baseline and 3 months
  24h ambulatory blood pressure

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events v4.0 | weeks 2, 4, 6, 8, 10, and 12
  Safety and tolerability of the intervention
Change in blood cellular NAD+ metabolism | baseline and 3 months
  Assessment of the "NAD+ metabolome" in circulating PBMCs

CONTACTS AND LOCATIONS:
Overall Officials: Michel Chonchol, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UColorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh ES, Opoku G, Darvish S, Craighead DH, Ostrow A, Rossman MJ, Steele CN, Struemph T, You Z, Seals DR, Chonchol M, Nowak KL. Sex Differences in Dementia and Mild Cognitive Impairment in Nondialysis CKD. Clin J Am Soc Nephrol. 2025 Nov 20. doi: 10.2215/CJN.0000000922. Online ahead of print. No abstract available. PMID 41264372